CLINICAL TRIAL: NCT05294380
Title: Determination of Sarcopenia Risk and Related Factors in Pediatric Oncological Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, FİLİZ TUNA, Assoc Prof, Trakya University
Other Study IDs: TÜTF-BAEK 2021/389
Record Dates: First submitted 2022-02-22; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Sarcopenia; Pediatric Cancer
Keywords: sarcopenia; Smartphone Addiction; Pediatric Cancer; Hematologic Malignancy; Anxiety Depression; bioelectrical impedance analysis
MeSH Terms: conditions — Sarcopenia; Neoplasms; Internet Addiction Disorder; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- oncologic: Be between the ages of 2-18 years Being under pediatric oncology outpatient/clinical follow-up Being able to stand unaided without using a cane/walker Exclusion criteria; Having any of the diagnoses of hypertension, any cardiac arrhythmia-conduction disorders, coronary artery disease, heart failure, diabetes mellitus, hyperlipidemia, cardiovascular diseases, COPD, pulmonary infection, active infection.
  Depression Illness that causes balance problems Peripheral vascular disease Presence of disease that prevents standing up with support Presence of diseases that may cause muscle mass loss (cerebral palsy, neuromuscular disease, congenital metabolic disorder, brain damage) mental retardation Children with a severe emotional disorder, adjustment disorder Physical disability to prevent safe and appropriate testing Having used anti-flu medicine in the last 1 week Failure to obtain consent
- control: Be between the ages of 2-18 years Exclusion criteria; Having any of the diagnoses of hypertension, any cardiac arrhythmia-conduction disorders, coronary artery disease, heart failure, diabetes mellitus, hyperlipidemia, cardiovascular diseases, COPD, pulmonary infection, active infection.
  Depression Illness that causes balance problems Peripheral vascular disease Presence of disease that prevents standing up with support Presence of diseases that may cause muscle mass loss (cerebral palsy, neuromuscular disease, congenital metabolic disorder, brain damage) mental retardation Children with a severe emotional disorder, adjustment disorder Physical disability to prevent safe and appropriate testing Having used anti-flu medicine in the last 1 week Failure to obtain consent

SUMMARY:
In children, both malnutrition and sarcopenia are associated with prolongation of hospital stay, increased morbidity, mortality, and health-related complications. While the decrease in muscle strength refers to "probable sarcopenia", "sarcopenia" is confirmed by adding the decrease in muscle quantity/quality to this situation. In case all three criteria are together, "severe sarcopenia" is mentioned. The aim of this study is the evaluate whether there is a difference in the risk of sarcopenia and related factors in pediatric oncological children compared to healthy controls matched for body mass index group, physical activity level group, sex, and age.

Our research was planned as cross-sectional and descriptive research. Patients diagnosed with pediatric oncologic cancer will be included. Demographic data, malnutrition, the risk for sarcopenia, physical activity status, smartphone addiction, fatigue, and hospital anxiety and depression will be evaluated with questionnaires.

Muscle strength (manual muscle strength assessment), Muscle quantity (the bilateral calf circumference with a tape measure and by bioelectrical impedance analysis (BIA)), and physical performance (Short Physical Performance Battery) will be evaluated by the physiotherapist.

The data of the research will be evaluated with the SPSS package program. After examining the conformity of the data that can be measured in statistical evaluations to a normal distribution with a single sample Kolmogorov Smirnov test, one-way analysis of variance will be applied for comparisons between groups for those with normal distribution, and t-test for independent groups. Kruskal Wallis analysis of variance and Mann Whitney U test will be used in the evaluation of data that do not conform to the normal distribution. Pearson χ2 and Yates corrected Pearson χ2 test Fisher's exact χ2 will be used for qualitative data. As descriptive statistics, numbers and percentages will be given for categorical data, and Median (Min-Max) values and arithmetic mean±standard deviation will be given for quantitative data. For all statistics, the limit of significance will be chosen as bidirectional p<0.05.

DETAILED DESCRIPTION:
As incidence and survival, rates increase in childhood and adolescent cancers, the importance of rehabilitation in this area increases (1-5). Functional limitations in the physical and cognitive domains are reported by children throughout the continuum of cancer care. These limitations are also experienced in very young children under 4 years of age with leukemia and lymphoma, adolescents and young adults struggling with leukemia, sarcoma, or central nervous system tumors (3, 6). Studies in adults who have won the childhood malignancy struggle report adulthood problems. Among these problems, deterioration of physical function, decrease in physical fitness, deterioration of neurocognition, fatigue, and pain, which affect their employment, participation in the life, and quality of life, are reported (2, 5, 7, 8). The roles of rehabilitation professionals, physical medicine and rehabilitation specialists, and physiotherapists in the childhood cancer population are particularly emphasized in the literature to prevent these limitations (1).

Malnutrition in children with chronic diseases is a common condition that causes problems in patient care. Sarcopenia or decreased musculoskeletal muscle mass contributes to the alteration of muscle function. This has been demonstrated in adults with chronic disease, but its impact on clinical outcomes in children has not been adequately described in the pediatric literature. Research in this area is affected by the lack of a uniform definition of sarcopenia in children. However, there is concern that childhood sarcopenia may have a long-term negative impact on growth, neurocognitive development, and quality of life-extending into adulthood. The similarities between sarcopenia and malnutrition are depleted lean muscle mass, changes in muscle function, and suboptimal food intake leading to nutritional deficiencies. In pediatric patients, this leads to growth failure and a potential neurodevelopmental delay in cognition, gross and fine motor development.

In children, both malnutrition and sarcopenia are associated with prolongation of hospital stay, increased morbidity, mortality, and health-related complications (3).

In adult oncological patients (over 18 years of age), the risk of sarcopenia, which is stated to predict malnutrition, is reported to be 40% (9).

As the investigators mentioned before, there is no single definition of sarcopenia with strict rules in childhood sarcopenia. However, in the 2019 European update, three criteria are emphasized in the diagnosis of sarcopenia for elderly individuals. These criteria are:

* decrease in muscle strength,
* decrease in muscle quantity or quality, and
* is stated as a decrease in physical performance. While the decrease in muscle strength refers to "probable sarcopenia", "sarcopenia" is confirmed by adding the decrease in muscle quantity/quality to this situation. In case all three criteria are together, "severe sarcopenia" is mentioned. The same update raises "red flags" in screening for sarcopenia. These red flags include: general weakness, visual loss of muscle mass, decreased muscle strength of the arms or legs, slow walking speed, fatigue, falls, loss of weight, loss of energy, and difficulty performing activities of daily living (10). Therefore, current research aims to question these criteria and the existence of red flags in the pediatric population.

Whether a sedentary lifestyle or physical inactivity due to the disease contributes to the development of sarcopenia (11).

Smartphone addiction is suggested as one of the causes of physical inactivity. Therefore, our study, it is aimed to evaluate both situations.

Physical fitness is the ability to correctly and successfully perform occupational, recreational, and daily activities without fatigue.

It includes two main components: health-related physical fitness (body composition, cardiorespiratory endurance, muscle strength and endurance, flexibility) and performance-related physical fitness (balance, coordination, reaction time, agility, speed, and power). In the current study, pediatric oncology will be evaluated in both patient and control participants.

In future directions for body composition assessments in pediatric oncological cases, "determining the prevalence and clinical significance of sarcopenia and sarcopenic obesity, which are potentially modifiable risk factors, will improve current understanding of the patient's nutritional status, assist in the early identification of those at greatest risk for adverse outcomes, and assist clinicians in their treatment plans. It will enable them to optimize and improve their effects" (12). Further research in this area could lead to improving and customizing chemotherapy dose, optimizing the timing of nutritional and physiotherapy supportive care interventions, and increasing tolerance to both traditional and new treatments. Therefore, progress in this area may have a long-term impact on the patient's quality of life and successful transition to survival (13).

Purpose of the research:

It aims to answer the question of whether there is a difference in the risk of sarcopenia and related factors in pediatric oncological children compared to healthy controls matched for body mass index group, physical activity level group, sex, and age.

Benefits and contributions of the research to science and society:

In the light of the information obtained as a result of the research, a window of opportunity will be provided for the rehabilitation service for the prevention of possible complications that may develop based on the sarcopenia status and related factors in pediatric oncological children, and it is anticipated that this will benefit science and the society.

Current research was planned as cross-sectional and descriptive research. Patients diagnosed with pediatric oncologic cancer will be included. Demographic data, malnutrition, the risk for sarcopenia, physical activity status, smartphone addiction, fatigue, and hospital anxiety and depression will be evaluated with questionnaires.

Muscle strength (manual muscle strength assessment), Muscle quantity (the bilateral calf circumference with a tape measure and by bioelectrical impedance analysis (BIA)), and physical performance (Short Physical Performance Battery) will be evaluated by the physiotherapist.

The data of the research will be evaluated with the SPSS package program. After examining the conformity of the data that can be measured in statistical evaluations to a normal distribution with a single sample Kolmogorov Smirnov test, one-way analysis of variance will be applied for comparisons between groups for those with normal distribution, and t-test for independent groups. Kruskal Wallis analysis of variance and Mann Whitney U test will be used in the evaluation of data that do not conform to the normal distribution. Pearson χ2 and Yates corrected Pearson χ2 test Fisher's exact χ2 will be used for qualitative data. As descriptive statistics, numbers and percentages will be given for categorical data, and Median (Min-Max) values and arithmetic mean±standard deviation will be given for quantitative data. For all statistics, the limit of significance will be chosen as bidirectional p<0.05.

When the literature on the subject of our study was examined, in the study of Lurz et al., computed tomography images of children aged 0-18 were compared by reviewing healthy pediatric trauma victims. In this retrospective study, 23 patients and 46 healthy controls were included. Considering this study and since it was calculated that 26 patients from each group should be included in the power analysis, in our study where muscle strength, muscle quantity/quality, and physical performance parameters will be compared, 30 patients between the ages of 2-18 with and without the pediatric oncological disease (probable case It is planned to include the child (taking into account the losses of the child).

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 2-18 years
* Being under pediatric oncology outpatient/clinical follow-up
* Being able to stand unaided without using a cane/walker

Exclusion Criteria:

* Having any of the diagnoses of hypertension, any cardiac arrhythmia-conduction disorders, coronary artery disease, heart failure, diabetes mellitus, hyperlipidemia, cardiovascular diseases, COPD, pulmonary infection, active infection.
* Depression Illness that causes balance problems
* Peripheral vascular disease
* Presence of disease that prevents standing up with support.
* Presence of diseases that may cause muscle mass loss (cerebral palsy, neuromuscular disease, congenital metabolic disorder, brain damage) mental retardation
* Children with a severe emotional disorder, adjustment disorder
* Physical disability to prevent safe and appropriate testing
* Having used anti-flu medicine in the last 1 week
* Failure to obtain consent.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants, who meet inclusion and exclusion criteria, with ages between 2 and 18 years will be selected from Trakya University Faculty of Medicine Pediatric Oncology outpatient polyclinic and clinic and Physical Therapy and Rehabilitation polyclinic and clinic.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-09-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Muscle quantity. | Seven months
  Bioelectrical impedance analysis (BIA) has been explored for estimation of total or Appendicular Skeletal Muscle Mass (ASM). BIA equipment does not measure muscle mass directly, but instead derives an estimate of muscle mass based on whole-body electrical conductivity. BIA uses a conversion equation that is calibrated with a reference of DXA-measured lean mass in a specific population. BIA equipment is affordable, widely available, and portable, especially single-frequency instruments. Muscle quantity will be determined by measuring the bilateral calf circumference with a tape measure and by BIA, which is considered one of the main standard tools for sarcopenia case-finding in clinical practice. Whole-body skeletal muscle mass (SMM) or Appendicular skeletal muscle mass (ASMM) predicted by BIA.
Physical performance | Seven months
  Physical performance will be determined by Short Physical Performance Battery (SPPB). The SPPB is a composite test that includes assessment of gait speed, a balance test, and a chair stand test.
Muscle strength. | Seven months
  Upper extremities (manual muscle strength assessment), the lower extremities will be evaluated (by manual muscle strength assessment and chair rise test). The chair stand test (also called chair rise test) can be used as a proxy for strength of leg muscles (quadriceps muscle group). The chair stand test measures the amount of time needed for a patient to rise five times from a seated position without using his or her arms; the timed chair stand test is a variation that counts how many times a patient can rise and sit in the chair over a 30-second interval. Since the chair stand test requires both strength and endurance, this test is a qualified but convenient measure of strength.

SECONDARY OUTCOMES:
Symptoms or signs of sarcopenia | Seven months
  "Red flags of sarcopenia" with a "family-oriented questionnaire"
The presence of malnutrition | Seven months
  The presence of malnutrition will be evaluated with the Simple Pediatric Nutrition Screening questionnaire.
Physical activity for parent | Seven months
  • Short Form International Physical Activity Questionnaire for Parent
Physical activity for preschool children and school-age children and adolescents | Seven months
  • Physical activity for preschool children and school-age children and adolescents
Physical activity for elementary 4-8th grades | Seven months
  • Physical activity scale (elementary 4-8th grades)
Smartphone Addiction | Seven months
  Smartphone Addiction (Parent and Child Smartphone Addiction Scale Short Form). The cut-off point is 29.5 for the Smartphone Addiction Scale-Short Version. When the score is greater than 29.50, the participant is determined as smartphone-addicted.
Childhood cancer fatigue | Seven months
  -Childhood cancer fatigue scale administered to mothers (• Child fatigue scale parent form (weekly)) The minimum and maximum scores are 17 and 85, respectively. An increase in score indicates an increase in fatigue.
Depression status | Seven months
  Depression status will be assessed with the Hospital Anxiety and Depression (HAD) Scale. The cut-off point is 10 for the anxiety subscale and 7 for the depression subscale.

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University Medical Faculty, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tanner L, Keppner K, Lesmeister D, Lyons K, Rock K, Sparrow J. Cancer Rehabilitation in the Pediatric and Adolescent/Young Adult Population. Semin Oncol Nurs. 2020 Feb;36(1):150984. doi: 10.1016/j.soncn.2019.150984. Epub 2020 Jan 24. PMID 31983485
- [Background] Fernandez-Pineda I, Hudson MM, Pappo AS, Bishop MW, Klosky JL, Brinkman TM, Srivastava DK, Neel MD, Rao BN, Davidoff AM, Krull KR, Mulrooney DA, Robison LL, Ness KK. Long-term functional outcomes and quality of life in adult survivors of childhood extremity sarcomas: a report from the St. Jude Lifetime Cohort Study. J Cancer Surviv. 2017 Feb;11(1):1-12. doi: 10.1007/s11764-016-0556-1. Epub 2016 Jun 4. PMID 27262580
- [Background] Ooi PH, Thompson-Hodgetts S, Pritchard-Wiart L, Gilmour SM, Mager DR. Pediatric Sarcopenia: A Paradigm in the Overall Definition of Malnutrition in Children? JPEN J Parenter Enteral Nutr. 2020 Mar;44(3):407-418. doi: 10.1002/jpen.1681. Epub 2019 Jul 22. PMID 31328301
- [Background] Phillips SM, Padgett LS, Leisenring WM, Stratton KK, Bishop K, Krull KR, Alfano CM, Gibson TM, de Moor JS, Hartigan DB, Armstrong GT, Robison LL, Rowland JH, Oeffinger KC, Mariotto AB. Survivors of childhood cancer in the United States: prevalence and burden of morbidity. Cancer Epidemiol Biomarkers Prev. 2015 Apr;24(4):653-63. doi: 10.1158/1055-9965.EPI-14-1418. PMID 25834148
- [Background] Ehrhardt MJ, Sandlund JT, Zhang N, Liu W, Ness KK, Bhakta N, Chemaitilly W, Krull KR, Brinkman TM, Crom DB, Kun L, Kaste SC, Armstrong GT, Green DM, Srivastava K, Robison LL, Hudson MM, Mulrooney DA. Late outcomes of adult survivors of childhood non-Hodgkin lymphoma: A report from the St. Jude Lifetime Cohort Study. Pediatr Blood Cancer. 2017 Jun;64(6):10.1002/pbc.26338. doi: 10.1002/pbc.26338. Epub 2016 Nov 15. PMID 27860222
- [Background] Kesting SV, Gotte M, Seidel CC, Rosenbaum D, Boos J. Motor Performance After Treatment for Pediatric Bone Tumors. J Pediatr Hematol Oncol. 2015 Oct;37(7):509-14. doi: 10.1097/MPH.0000000000000396. PMID 26207777
- [Background] Hudson MM, Oeffinger KC, Jones K, Brinkman TM, Krull KR, Mulrooney DA, Mertens A, Castellino SM, Casillas J, Gurney JG, Nathan PC, Leisenring W, Robison LL, Ness KK. Age-dependent changes in health status in the Childhood Cancer Survivor cohort. J Clin Oncol. 2015 Feb 10;33(5):479-91. doi: 10.1200/JCO.2014.57.4863. Epub 2014 Dec 29. PMID 25547510
- [Background] Ness KK, DeLany JP, Kaste SC, Mulrooney DA, Pui CH, Chemaitilly W, Karlage RE, Lanctot JQ, Howell CR, Lu L, Srivastava DK, Robison LL, Hudson MM. Energy balance and fitness in adult survivors of childhood acute lymphoblastic leukemia. Blood. 2015 May 28;125(22):3411-9. doi: 10.1182/blood-2015-01-621680. Epub 2015 Mar 26. PMID 25814529
- [Background] Borges TC, Gomes TLN, Pimentel GD. Sarcopenia as a predictor of nutritional status and comorbidities in hospitalized patients with cancer: A cross-sectional study. Nutrition. 2020 May;73:110703. doi: 10.1016/j.nut.2019.110703. Epub 2019 Dec 14. PMID 32007693
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Mijnarends DM, Koster A, Schols JM, Meijers JM, Halfens RJ, Gudnason V, Eiriksdottir G, Siggeirsdottir K, Sigurdsson S, Jonsson PV, Meirelles O, Harris T. Physical activity and incidence of sarcopenia: the population-based AGES-Reykjavik Study. Age Ageing. 2016 Sep;45(5):614-20. doi: 10.1093/ageing/afw090. Epub 2016 May 17. PMID 27189729
- [Background] Yip C, Dinkel C, Mahajan A, Siddique M, Cook GJ, Goh V. Imaging body composition in cancer patients: visceral obesity, sarcopenia and sarcopenic obesity may impact on clinical outcome. Insights Imaging. 2015 Aug;6(4):489-97. doi: 10.1007/s13244-015-0414-0. Epub 2015 Jun 13. PMID 26070723
- [Background] Joffe L, Schadler KL, Shen W, Ladas EJ. Body Composition in Pediatric Solid Tumors: State of the Science and Future Directions. J Natl Cancer Inst Monogr. 2019 Sep 1;2019(54):144-148. doi: 10.1093/jncimonographs/lgz018. PMID 31532526